CLINICAL TRIAL: NCT04131010
Title: Digital Catheter Based Pancreatoscopy (SpyGlassDS) for the Management of Symptomatic Pancreatic Duct Stones in Selected Patients With Chronic Pancreatitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Evangelisches Krankenhaus Düsseldorf (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPYGlass DS
Record Dates: First submitted 2019-07-08; First posted 2019-10-18 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Pancreatitis, Calcific; Pancreatitis, Chronic
MeSH Terms: conditions — Pancreatitis, Calcific; Pancreatitis, Chronic

STUDY DESIGN:
Intervention Model Description: International prospective multicenter cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- SpyGlass Pancreatoscopy (Experimental): ERP with direct pancreatoscopy
  Interventions: Device: single operator video cholangioscopy

INTERVENTIONS:
Device: single operator video cholangioscopy — The technique provides digital imaging with a higher resolution and improved maneuverability compared to the legacy fiberoptic system. In addition, the working channel was enlarged to a diameter of 1.3 mm. Retrospective data showed an overall technical success rate for single-operator video pancreatoscopy (SOVP) guided treatment of pancreatic stones of 95%

SUMMARY:
Investigation of the efficacy and safety of digital catheter-based pancreatoscopy (DCP) for the Treatment of symptomatic Stones of the pancreatic duct in selected patients with chronic calcifying pancreatitis (CCP)

DETAILED DESCRIPTION:
Background Endoscopic treatment of patients with chronic calcifying pancreatitis (CCP) is still challenging and controversially discussed. The goal is symptom control and relief of pain, which can be achieved by draining an obstructed main pancreatic duct (MPD) and/or removal of ductal stones. The 2012 European Society of Gastrointestinal Endoscopy (ESGE)- Guidelines recommends ESWL as a first step for patients with uncomplicated painful chronic pancreatitis and radiopaque stones ≥5mm obstructing the MPD. However, limitations of ESWL (extracorporeal shockwave lithotripsy ) include its limited availability, a likely need for multiple sessions and often repeated ERCP (endoscopic retrograde cholangiopancreatography) sessions for removal of stone fragments or treatment of associated strictures.

Pancreatoscopically guided management of pancreatic stones offers a potential alternative to ESWL. However, the numbers of studies and enrolled patients are still low. In 2015 single operator video cholangioscopy (SpyGlassDS, Boston Scientific) was introduced. Available data on its use for pancreatoscopy is limited. The technique provides digital imaging with a higher resolution and improved maneuverability compared to the legacy fiberoptic system. In addition, the working channel was enlarged to a diameter of 1.3 mm. Although SOVP have shown promise in CCP, studies to date generally have been limited by: retrospective design, relatively small and mixed patient populations, short follow-up periods, different clinical and technical endpoints, and, often, a single-center design. Therefore, the investigators designed a prospective multicenter cohort study to evaluate long-term clinical efficacy, technical success and safety of SOVP.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients are adults (≥ 18 years of age) with a signed informed consent with:
* symptomatic chronic pancreatitis (recurrent pain attacks, history of pain for at least 3 months), and
* ≤3 radiopaque stones ≥5mm obstructing the MPD in the pancreatic head and/or corpus.

Exclusion Criteria:

* - Health status ASA 4
* Pregnancy
* Coagulopathy (INR≥2.0, Platelets < 70/nl)
* Taking anti-platelet agents or anticoagulants (other than aspirin) within last 7 days
* Any medical contraindication to ERCP, deep sedation or general anesthesia
* History of chronic symptomatic pancreatitis of more than 3-4 years[9]
* History of daily use of opioids except Tramadol for more than 6 months in the last 2 years
* Episode of biliary obstruction in the previous 2 months (defined as jaundice or bilirubin levels >=2,5mg/dl or CBD stent
* Auto-Immune Pancreatitis or IgG4 associated pancreatitis
* Altered GI anatomy, previous failures of endoscopic approach to the papilla
* Abdominal pain not attributable to CP
* Any suspicion of pancreatic cancer
* Current symptomatic WON
* More than one ductal stricture in the pancreatic head or body
* Previous ESWL pancreatic stones
* Age <18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2019-05-31 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with complete clearance of the MPD from ≤3 stones in the pancreatic head and/or body by means of SOVP in ≤3 treatment sessions | at baseline visit
  Number of patients where complete clearance of the MPD could be reached within three Treatment sessions of SOVP

SECONDARY OUTCOMES:
Number of treatment sessions | within three months
  Number of Treatment sessions which are necessary to reach complete clearanceof the MPD
Procedural time | at baseline visit
  Time for the procedure from beginning to the end of the intervention
Number of participants with Adverse events (post procedure and at 30 days) | at baseline visit and 30 days after the invention
  Incidence of Treatment-emergent Adverse Events as reported by the patients or as detected during the visits or by unplanned hospitalization
Rate of pancreatoscopic visualization of the targeted stones(s) and initiation of lithotripsy by using the Single-Operator Video pancreatoscopy (SOVP) | at baseline visit
  Determined by number of patients where the targeted Stones can be made visuable during the intervention
Number of patients with stone fragmentation (particles ≤3mm, or decreased stone density at X-ray, an increased stone surface and heterogenity of the stone(s) which may fill the MPD and adjacent side branches | at baseline visit
  Number of patients where the Stones can be fragmented during the intervention
Number of patients with ductal drainage after complete or incomplete ductal clearance (e.g. by placement of an endoprosthesis) | at baseline visit
Determination by MRCP of the diameter of the MPD prior to treatment and at 6 months after the final intervention | prior procedure and 6 months after procedure
Rate of patients with improved Clinical Outcome or complications as assessed by Numeric Rating scale (NRS) for pain, Izbicki Pain Score and number of pain attacks determined at 30 days, 6 and 12 months after the final intervention by means of SOVP | 30 days, 6 months and 12 months after procedure
  Self-reported pain Status as assessed by the pain assessments NRS for pain and Izbicki pain Score as well as self-reported pain attacks
Change of Quality of life as assessed by the Short Form -12 questionnaire prior to treatment and 6 months after the final intervention | prior treatrment, 6 months after treatment and at the last procedure visit (procedure I, II or III as applicable)
  Self-reported Quality of life as assessed by the Short Form -12 questionnaire (this questionnaire is evaluated centrally by the rights-holding company), answering 12 questions regarding Quality of Life

CONTACTS AND LOCATIONS:
Locations (1):
- Evangelisches Krankenhaus Düsseldorf, Düsseldorf, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No